CLINICAL TRIAL: NCT04896645
Title: Albuterol Integrated Adherence Monitoring in Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Neema Izadi, Assistant Professor, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-20-00013
Record Dates: First submitted 2021-05-12; First posted 2021-05-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients 8 to <19 years of age with a diagnosis of asthma (Experimental): Patients 8 to <19 years of age with a diagnosis of asthma as ICD-9 code 493 or ICD-10 code J45 seen in the allergy clinic at CHLA who have an albuterol rescue inhaler already prescribed and access to a personal smartphone will be eligible for recruitment.
  Interventions: Device: Digihaler Albuterol Device by TEVA

INTERVENTIONS:
Device: Digihaler Albuterol Device by TEVA — Patient with asthma will have their regular albuterol rescue inhaler replaced with Digihaler, they will also be asked to perform gamified spirometry (Aluna) at home
  Other Names: Electronic Adherence Monitor

SUMMARY:
The investigators propose to evaluate whether an integrated electronic adherence monitoring albuterol rescue inhaler can improve proper use in a mostly minority and inner-city population of children treated for asthma at the Children's Hospital of Los Angeles

DETAILED DESCRIPTION:
This study is designed to (1) determine whether an integrated EAM albuterol rescue inhaler can increase proper use (2) determine if the monitoring capabilities of the device (flow rate, warnings) and/or increased proper use from having the device correlate with better outcomes. The investigators will also have patients perform at-home gamified spirometry (Aluna ©) to (3) determine if at-home spirometry can predict albuterol use or change outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 8 to <19 years of age with a diagnosis of asthma as ICD-9 code 493 or ICD-10 code J45 seen in the allergy clinic at CHLA who have an albuterol rescue inhaler already prescribed and access to a personal smartphone will be eligible for recruitment.

Exclusion Criteria:

* Patients unable to use device, unable to use albuterol (i.e. must use levalbuterol) or Age < 4 (ProAir® Digihaler only approved for Subjects 4 years and older). Patients with other chronic lung disease besides asthma or other significant comorbidities that could affect lung function/asthma (e.g. significant heart defects, immunodeficiency, cystic fibrosis, etc).

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Asthma Outcomes | 3 months
  Severity by NHLBI EPR3 Guidelines
Asthma Adherence | 3 months
  4-item Morisky Medication Adherence Scale (MMAS-4)
Asthma Adherence | 3 months
  Test of Adherence to Inhalers (TAI)
Asthma Outcomes | 3 months
  Composite Asthma Severity Index (CASI)
Asthma Outcomes | 3 months
  Asthma Control Test (ACT)
Albuterol Use | 3 months
  Questionnaires created by investigators addressing when and how often albuterol is used for symptoms, illness, etc.

SECONDARY OUTCOMES:
Spirometry | 3 months
  Aluna at home gamified spirometer, measures full spirometry FEV1, FVC, FEV1/FVC, Peak Flow.
Lung Function | 3 months
  Microlife FEV1, measures FEV1
Asthma Quality of Life | 3 months
  PedsQL (Pediatric Quality of Life Inventory)

CONTACTS AND LOCATIONS:
Overall Officials: Neema Izadi, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No